CLINICAL TRIAL: NCT05871788
Title: Biomarkers in Patients With Metastatic Breast Cancer
Acronym: BIOPEACE
Status: Not yet recruiting | Type: Observational
Sponsor: Tunisian Association for Immuno-oncology Research (Other)
Responsible Party: Sponsor
Other Study IDs: ECOCS2020-01
Record Dates: First submitted 2023-05-13; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Identify the Number of Eligible Patients for Immunotherapy According to the Epidemiological and Biological Profile in Tunisia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — blood sample, biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: identify biomarkers — Identify the epidemiological profile of the biological signature (PD-L1 / TMB / MSI/HRD/ TILs) of patients with locally advanced or metastatic breast carcinoma

SUMMARY:
In order to allow Tunisian patients with breast cancer to access immunotherapies, and innovative treatments to extend life expectancy of patients with breast cancer with a poor prognosis, it is important to study the epidemiological profile of Tunisian cancers breast, in terms of PD-L1 expression, tumor mutational burden (TMB), microsatellite instability status (MSI) and rate of TILs, in metastatic and locally advanced cases, in Tunis, over a one-year follow-up period.

It is also important to study other inflammatory and tumor biomarkers which would have a prognostic or even therapeutic value:

* serum dosage of LDH (lactate dehydrogenase)
* IL-6 (interleukin 6)
* CRP (C-reactive protein)
* absolute count of lymphocytes (CLA) and eosinophils
* quantification of circulating tumor DNA before treatment and under treatment. The primary objective id to identify the epidemiological profile of the biological signature (PD-L1 / TMB / MSI/HRD/ TILs) of patients with locally advanced or metastatic breast carcinoma before and during the systemic treatment.

DETAILED DESCRIPTION:
Procedure:

1. Verification of the inclusion / non-inclusion criteria
2. Signing the consent form
3. Surgical, Medical and family history, ongoing treatments
4. Clinical Examination1
5. Radiological examinations 2
6. TNM Classification (Appendix 3)
7. Standard biochemical assessment 3
8. Inflammatory assessment (CRP, LDH, IL6)
9. Hematological assessment (NFS, platelets)
10. Tumor markers (ACE, CA15-3)
11. Histological and molecular examination 4:

    * Expression PD-L1 by IHC (Immuno-Histochemistry)
    * TILs by IHC
    * - MSI status: MMR * proteins (Mismatch Repair Protein) (Appendix 4) by NGS via TruSight™ Oncology 500 Kit (Illumina) , if PD-L1>1%
    * Score HRD : by NGS via TruSight™ Oncology 500 Kit (Illumina) , if PD-L1>1%
    * TMB mutational burden by next generation sequencing "Next Generation Sequencing" (NGS) via TruSight™ Oncology 500 Kit (Illumina) if PD-L1>1%
    * tDNA by digital PCR
12. Radiological evaluation5
13. Indication of surgery? (if yes type of surgery to be specified)
14. Evaluation of adverse events / effects: Tolerance of the previous treatment
15. Completion the source documents and the eCRF

    Clinical Exam1:
    * General State according to the WHO classification or according to the Karnowsky Index
    * Breast examination: inspection (symmetry, appearance of the skin), palpation (size of the tumor, presence of mammary discharge).
    * Examination of the axillary and supraclavicular lymph node areas
    * Abdominal examination
    * Pulmonary auscultation
    * Skeleton examination Radiological examination2:
    * Mammography and echo-mammary
    * Thoraco-abdomino-pelvic CT scan
    * Bone scintigraphy
    * Cardiac ultrasound

    Standard biochemical balance3:

    Blood group, creatininemia, blood ionogram, calcemia, glycemia, bilirubin, transaminases, gamma-GT, alkaline phosphatases, total cholesterol, triglycerides, uric acid, albuminemia.

    Histological examination4:
    * Biopsy with part number assigned by the laboratory, name of the laboratory
    * Histological type
    * Grade of Scarff-Bloom and Richardson (SBR)
    * Estrogen receptors, progesterone receptors
    * Her2Neu
    * Ki67
    * PD-L1
    * TILs
    * MMR

    Molecular Examination4:
    * MSI status by pentaplex PCR and capillary electrophoresis by NGS platform via the TruSight™ kit Oncology 500 (Illumina)
    * HRD Score by NGS platform via the TruSight™ kit Oncology 500 (Illumina)
    * Mutational burden TMB by NGS platform via the TruSight™ kit Oncology 500 (Illumina)
    * Circulating tumor DNA by digital PCR Radiological assessment5:
    * If the stage is locally advanced (appendix 3): Breast ultrasound +/- Mammography +/- Breast MRI
    * If metastatic stage: Thoraco-abdomino-pelvic CT scan 12 | 27 Visit details

      • Initial visit D0 (V1)
      * Signature of informed consent form
      * Verification of inclusion / non-inclusion criteria
      * Medical, surgical and family history
      * Current treatments
      * Clinical examination1
      * Radiological examinations2
      * TNM classification
      * Standard biochemical assessment3
      * Inflammatory assessment (CRP, LDH, IL6)
      * Hematological assessment (NFS, platelets)
      * Tumor markers (ACE, CA15-3)
      * Histological examination with immunohistochemistry and molecular4:
    * Biopsy with part number assigned by the lab, name of the lab
    * Histological type
    * SBR grade
    * Estrogen receptors, progesterone receptors
    * Her2Neu
    * Ki67
    * PD-L1
    * TILs
    * MMR
    * MSI
    * HRD
    * TMB mutational charge
    * ctDNA o Completion of source documents and eCRF

      * Visit after 3 chemotherapy treatment cycles (V2)

        * Current treatments
        * Clinical examination1
        * Hematological assessment (NFS, platelets)
        * Tumor markers (ACE, CA15-3)
        * Radiological assessment5
        * Evaluation of adverse events / effects: Tolerance of the previous treatment
        * Completion of source documents and eCRF
      * Assessment visit (V3) o Current treatments

        o Clinical examination1
        * TNM classification
        * Inflammatory assessment (CRP, LDH, IL6)
        * Hematological assessment (NFS, platelets)
        * Tumor markers (ACE, CA15-3)
        * Histological examination with immunohistochemistry and molecular4:
    * Biopsy with part number assigned by the lab, name of the lab
    * Histological type
    * SBR grade 13 | 27
    * Estrogen receptors, progesterone receptors
    * Her2Neu
    * Ki67
    * PD-L1
    * TILs
    * ctDNA

      o Radiological assessment5

      o Assessment of adverse events / effects

      o Fill in the source files and the eCRF
      * Follow-up visit at 3 months (V4)

        o Current treatments

        o Clinical examination1

        o Tumor markers (ACE, CA15-3)

        o Radiological examinations2

        o Evaluation of adverse events / effects
        * Completion of source documents and eCRF
      * Follow-up visit at 6 months (V5) o Current treatments o Clinical examination1 o Tumor markers (ACE, CA15-3)

        * Radiological examinations2
        * Evaluation of adverse events / effects
        * Completion of source documents and eCRF

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Signed informed consent
* Histological evidence of breast carcinoma.
* Locally advanced (stage III inoperable) or metastatic (stage IV) carcinoma, the metastases of which have been diagnosed straight away or after adjuvant or neoadjuvant treatment.
* No treatment for metastatic disease.
* Metastatic disease: histological evidence of metastasis
* Patients who will receive systemic treatment (chemotherapy, targeted therapy, hormone therapy)
* Life expectancy greater than 3 months

Exclusion Criteria:

* Non-epithelial breast cancer
* Non-biopsiable metastases
* Patients who have received before systemic treatment for metastatic disease (chemotherapy, targeted therapy, hormone therapy)
* Patients with a contraindication to chemotherapy, and / or hormone therapy, and

  / or targeted therapy.
* Foreign patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with metastatic or locally advanced breast cancer in Tunis, Tunisia.
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
number of eligible patients for immunotherapy | 2023 to 2027
  Identify the number of eligible patients for immunotherapy according to the epidemiological and biological profile

SECONDARY OUTCOMES:
Relevance of immunotherapy in Tunisia | 2023 to 2027
  Assess the relevance of the introduction of immunotherapy in Tunisia, by calculating the extension of the life expectancy (without disease and overall) of the patients who could benefit from this treatment, compared to the cost.
  - Identify the sub-population of patients who benefit most from immunotherapy in Tunisia

IPD SHARING:
Plan to Share IPD: Undecided